CLINICAL TRIAL: NCT05927948
Title: Evaluating the Safety and Efficacy of Laight®-Therapy Treatment in Subjects With Hidradenitis Suppurativa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB11922
Record Dates: First submitted 2019-03-26; First posted 2023-07-03 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: The patient has one side exposed to treatment and the other side receives no treatment as the comparison. Hence, patient serves as their own control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): This is a split body study. The patients will serve as their own control. The side that receives Laight therapy will be randomized. For example, if the patient receives Laight therapy on the right, then the control will be the left.
  Interventions: Device: Laight therapy, NICE V3.1 device
- Control (No Intervention): This is a split body study. The patients will serve as their own control. The control side of the body will be randomized. For example, if the patient receives Laight therapy on the right, then the control will be the left.

INTERVENTIONS:
Device: Laight therapy, NICE V3.1 device — Laight therapy is a non-invasive method of treatment for HS and acne developed in Germany which utilizes a combination of radiofrequency and intense pulsed light exposure. Three passes of the device, all coupled with radiofrequency, are used in the proposed treatment area. The first pass encompasses wavelengths between 420 nm and 1200 nm, the second between 510 nm and 1200 nm, and the third pass between 690 nm and 1200 nm.
  Arms: Intervention

SUMMARY:
Hidradenitis suppurativa (HS) is a debilitating and chronic condition characterized by recurrent episodes of inflammation associated with the formation of abscesses, inflammatory nodules, pain, and drainage ultimately culminating in the formation of scarring in moderate to severe disease. HS affects more women than men in a ratio of approximately 3:1, and onset of the disease is typically after puberty. The axillae, breasts, groin, buttocks, and lower abdomen are common intertriginous regions which are affected by HS, and significant impacts on quality of life are reported in the literature.

The Hurley Staging system is commonly utilized to classify the severity of a patient's hidradenitis suppurativa. Stage 1 disease consists of one or more abscesses with no sinus tract formation or scarring. Stage 2 disease involves one or more widely separated recurrent abscesses, with formation of a sinus tract and/or scarring. Stage 3 involves multiple interconnected sinus tracts and/or abscesses throughout an anatomical area.

Histologic studies of HS suggest that follicular hyperkeratosis and obstruction is the primary event in the pathogenesis. Subsequently, there is rupture of the follicular infundibulum and a resulting inflammatory cascade. Despite recurrent episodes of purulent drainage, bacteria do not appear to play a primary role in the pathogenesis.

The traditional repertoire of treatment options for HS can be divided into medical and surgical options, however there is currently no cure for HS and treatments focus on symptomatic control. Medical treatments including topical and systemic antibiotics, hormonal agents, and biologic medications can successfully control symptoms however discontinuation of many of these is associated with relapses in disease symptoms. Conversely, surgical interventions such as traditional surgical excision performed in an operating room, or carbon dioxide laser excision performed under local anesthetic in an outpatient setting can induce long term symptom control however may not be appropriate for all patients considering the risk of general anesthesia, high cost of inpatient hospitalizations, and cumbersome healing process for procedures which heal by secondary intention. Despite numerous treatment options for HS, efficacious and non-invasive treatment options which result in long term remission of disease are needed to meet the needs of HS patients.

DETAILED DESCRIPTION:
Subjects receive treatment every 2 weeks for a total of 22 weeks, 10 treatments. Subject treatment side will be randomized via computer generated assignments.

Ultrasound imaging will be utilized to assess abscesses, nodules, and sinus tracts at investigator discretion. Patient-reported outcome measures include DLQI and Pain VAS. Physician-reported outcome measures include: HS-PGA, IHS4, Hurley Staging, and HiSCR.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old.
2. Have a diagnosis of Hurley stage I or II HS.
3. Patients must have bilateral HS in the axilla, groin, or breast.
4. Hurley stage 1 or 2 disease in either the axillae, groin, or inframammary locations.
5. At least 2 clinically observable lesions in the axilla, groin or breast.
6. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form.
7. Agree to follow and undergo all study-related procedures.

Exclusion Criteria:

1. No diagnosis of HS in the axillae or groin.
2. Tattoos located on proposed treatment locations.
3. Metal implants of intended treatment areas.
4. History of acne conglobata.
5. Concomitant use of antibiotics in the tetracycline class or oral or topical retinoids (permitted with 14-day washout period).
6. Concomitant use of biologic medications (6-month washout period).
7. Concomitant use of other topical treatments of HS in intended treatment locations (14-day washout period), except for topical benzoyl peroxide or topical clindamycin gel or lotion.
8. History of melanoma.
9. Active skin cancer in the proposed treatment area (non-melanoma in the past 6 month).
10. Current Nd:YAG laser hair removal for HS treatment in the study area.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Hurley Stage | 22 weeks
  Classification of HS severity Participant treatment location will be assessed using the Hurley Staging scale Stage I (Mild) Inflammatory nodule or abscess formation, single or multiple, without sinus tracts and scarring Stage II (Moderate) Recurrent abscesses and nodules with sinus tract formation or scarring: single or multiple widely separated lesions Stage III (Severe) Diffuse or near-diffuse involvement with multiple interconnected sinus tracts, scarring, and abscesses across entire area

SECONDARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response Score | baseline and end of treatment (22 weeks)
  Severity and activity of hidradenitis suppurativa assessment with a target of reaching a 50% reduction in the AN (abscess nodule) count
  HiSCR:
  * Abscesses: fluctuant, with or without drainage, tender or painful
  * Inflammatory nodules: tender, erythematous, pyogenic granuloma lesion
  * Draining fistulas: sinus tracts, with communications to skin surface, draining purulent fluid
    • Definition
  * AN (abcess nodule) Count= Abscess and inflammatory nodule count
  * At least a 50% reduction in AN count
  * No increase in the number of abscesses
  * No increase in the number of draining fistulas from baseline
Dermatology Life Quality Index | baseline and end of treatment (22 weeks)
  patient reported outcome measure of quality of life assessment
  DLQI Scoring SCORING
  The scoring of each question is as follows:
  Very much, scored 3 A lot scored, 2 A little scored, 1 Not at all scored, 0 Not relevant scored, 0 Question 7, 'prevented work or studying', scored 3 The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  DLQI SCORE INTERPRETATION 0 - 1 no effect at all on patient's life 2 - 5 small effect on patient's life 6 - 10 moderate effect on patient's life 11 - 20 very large effect on patient's life 21 - 30 extremely large effect on patient's life
Hidradenitis suppurativa physician global assessment | baseline and end of treatment (22 weeks)
  physician global assessment of HS severity
  HS PGA Clear 0 abscesses, 0 draining fistulas, 0 inflammatory nodules, and 0 noninflammatory nodules
  Minimal 0 abscesses, 0 draining fistulas, 0 inflammatory nodules, and presence of noninflammatory nodules
  Mild 0 abscesses, 0 draining fistulas, 1-4 inflammatory nodules Or 1 abscess or draining fistula and inflammatory nodules
  Moderate 0 abscesses, 0 draining fistulas, and ≥ 5 inflammatory nodules Or 1 abscess or draining fistula and ≥ 1 inflammatory nodule Or 2-5 abscesses or draining fistulas and < 10 inflammatory nodules
  Severe 2-5 abscesses or draining fistulas and ≥ 10 inflammatory nodules Very Severe >5 abscesses or draining fistulas
International HS Severity Scoring | baseline and end of treatment (22 weeks)
  severity scoring
  IHS4 (points)= Number of nodules x 1 + Number of abscesses x 2 + Number of draining tunnels (fistulae/sinuses) x 4
  A total score of 3 or less signifies mild, 4-10 signifies moderate and 11 or higher signifies severe disease.
Pain Visual Analog Scale | 22 weeks
  Scale of 1-10, 1 being the least amount of pain, 10 being the most amount of pain

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital Systems- New Center One, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tierney E, Mahmoud BH, Hexsel C, Ozog D, Hamzavi I. Randomized control trial for the treatment of hidradenitis suppurativa with a neodymium-doped yttrium aluminium garnet laser. Dermatol Surg. 2009 Aug;35(8):1188-98. doi: 10.1111/j.1524-4725.2009.01214.x. Epub 2009 May 12. PMID 19438670
- [Background] Wilden S, Friis M, Tuettenberg A, Staubach-Renz P, Wegner J, Grabbe S, von Stebut E. Combined treatment of hidradenitis suppurativa with intense pulsed light (IPL) and radiofrequency (RF). J Dermatolog Treat. 2021 Aug;32(5):530-537. doi: 10.1080/09546634.2019.1677842. Epub 2019 Oct 17. PMID 31609667